CLINICAL TRIAL: NCT02635984
Title: Randomized, Placebo Controlled Study of FOND (Fosaprepitant, Ondansetron, Dexamethasone) Versus FOND+O (FOND Plus Olanzapine) for the Prevention of Chemotherapy Induced Nausea and Vomiting in Hematology Patients Receiving Highly Emetogenic Chemotherapy Regimens
Brief Title: Study of FOND Versus FOND+O for the Prevention of CINV in Hematology Patients Receiving Highly Emetogenic Chemotherapy Regimens
Acronym: FOND-O
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Principal Investigator, Amber Clemmons, Pharmacist, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 818888
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Complications of Bone Marrow Transplant; Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triplet Therapy Plus Placebo (Placebo Comparator): All subjects will receive standard triplet antiemetic therapy which consists of ondansetron and dexamethasone on each day of chemotherapy plus fosaprepitant 150 mg IV once per national guidelines for CINV prophylaxis. In addition to those antiemetics, subjects will receive placebo on all chemotherapy days and for three additional days post chemotherapy.
  Interventions: Drug: Placebo
- Triplet Therapy Plus Olanzapine (Active Comparator): All subjects will receive standard triplet antiemetic therapy which consists of ondansetron and dexamethasone on each day of chemotherapy plus fosaprepitant 150 mg IV once per national guidelines for CINV prophylaxis. In addition to those antiemetics, subjects will receive olanzapine 10mg orally on all chemotherapy days and for three additional days post chemotherapy.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 10mg by mouth once daily on all chemotherapy days and for three days post-chemotherapy
  Other Names: Zyprexa
  Arms: Triplet Therapy Plus Olanzapine
Drug: Placebo — Placebo tablet taken by mouth once daily on chemotherapy days and for 3 days post chemotherapy
  Arms: Triplet Therapy Plus Placebo

SUMMARY:
The objective of this study is to compare the effectiveness of olanzapine added to standard triplet therapy (fosaprepitant, ondansetron, and dexamethasone) versus triplet therapy alone in preventing chemotherapy-induced nausea and vomiting (CINV) in hematology patients receiving highly or moderately emetogenic chemotherapy regimens.

DETAILED DESCRIPTION:
Nausea and vomiting remains a common and difficult to manage consequence of chemotherapy despite prophylaxis. These symptoms can often lead to a decreased quality of life, dehydration, and malnutrition. Olanzapine is an atypical antipsychotic that blocks multiple neuronal receptors involved in nausea/vomiting pathways. Olanzapine has been studied for breakthrough chemo-induced nausea and vomiting (CINV) as well as in prophylaxis of highly and moderately emetogenic regimens (HEC and MEC, respectively). However, these studies have focused on patients with solid tumor malignancies and chemotherapy regimens of short duration. To date, no publications have reported outcomes from adding olanzapine to standard triplet therapy, for hematology patients, including those undergoing hematopoietic stem cell transplants and those who receive multi-day HEC and MEC regimens.

This is a blinded, placebo controlled trial randomizing patients to receive olanzapine 10 mg orally on all chemotherapy days plus three additional days post chemotherapy or placebo in addition to standard triplet therapy (ondansetron and dexamethasone on each day of chemotherapy and fosaprepitant 150 mg IV on day one of chemotherapy). Inclusion criteria: age 18 or older, receiving inpatient or outpatient HEC or MEC chemotherapy including those regimens given before stem cell transplantation (ABVD, ICE ± R, 7+3 or 5+2, BEAM, Bu/Cy ± ATG, Bu/Flu ± ATG, FluCy ± ATG, BuMel, FluBuCy, Melphalan). Exclusion criteria: allergy to olanzapine, documented nausea/vomiting ≤24 hours before enrollment, treatment with other antipsychotic agents, or declined informed consent. Patients will be randomized to placebo or olanzapine in a block design stratified by chemotherapy type (transplant conditioning vs. chemotherapy only) and number of days of chemotherapy (single vs. multi-day) by the Investigational Drug Pharmacy services at Augusta University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient or outpatient hematology patient receiving one of the following regimens:
* Chemotherapy for hematologic malignancy:
* ABVD
* ICE ± R
* 7+3
* Conditioning therapy for stem cell transplantation:
* BEAM
* Bu/Cy ± ATG
* Bu/Flu ± ATG
* FluCy ± ATG
* FluCy + TBI
* BuMel
* FluBuCy
* Melphalan
* Etoposide + TBI
* Cyclophosphamide + TBI

Exclusion Criteria:

* Allergy to olanzapine
* Documented nausea or vomiting ≤24 hours prior to enrollment
* Treatment with other antipsychotic agents such as risperidone, quetiapine, clozapine, phenothiazine or butyrophenone ≤30 days prior to enrollment or planned during protocol therapy
* Chronic alcoholism
* Pregnant
* Declined or unable to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber B Clemmons, PharmD, Principal Investigator — Augusta University Medical Center
Locations (1):
- Augusta University Medical Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemmons AB, Orr J, Andrick B, Gandhi A, Sportes C, DeRemer D. Randomized, Placebo-Controlled, Phase III Trial of Fosaprepitant, Ondansetron, Dexamethasone (FOND) Versus FOND Plus Olanzapine (FOND-O) for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Patients with Hematologic Malignancies Receiving Highly Emetogenic Chemotherapy and Hematopoietic Cell Transplantation Regimens: The FOND-O Trial. Biol Blood Marrow Transplant. 2018 Oct;24(10):2065-2071. doi: 10.1016/j.bbmt.2018.06.005. Epub 2018 Jun 13. PMID 29906570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Started | 53 | 55
Completed | 50 | 51
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Study Arm Closed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Median (Full Range); unit: years] | 56 [22 to 74] | 54 [22 to 72] | 55 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 19 | 22 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 21 | 40
  White | 29 | 27 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Treatment Regimen [Count of Participants; unit: Participants]
  Chemotherapy Alone | 16 | 17 | 33
  HCT Conditioning | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Overall Percentage of Patients Who Had a Complete Response
Description: Overall percentage of patients who had a complete response (CR) defined as no emesis and minimal nausea (< 25 mm on a 100 mm visual analog scale [VAS]) during the overall assessment period (starting day 1 of chemotherapy and continuing for 5 days after discontinuation of chemotherapy) for the first cycle of chemotherapy.
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 13 | 28
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Based on an 80 % power and an alpha of 0.05, we estimated a need for 49 patients in each treatment arm. From a review of existing literature, the sample size was based on an estimated CR achieved in 65 % of patients on triplet therapy alone and a hypothesized clinically relevant increase of 25 % for the treatment group to 90 %; Test type: Superiority; p = 0.003, Chi-squared

2. Secondary Outcome: Percent of Patients With no Significant Nausea in Overall Assessment Period
Description: Reported for overall phases [chemotherapy days plus 5 days after] where all VAS < 25 mm
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 14 | 30
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Test type: Superiority; p = 0.001, Chi-squared

3. Secondary Outcome: Percent of Patients Achieving Complete Protection in Overall Assessment Phase
Description: (CP = no emesis, no breakthrough antiemetic use, no significant nausea). To be reported as overall phases [chemotherapy days plus 5 days after]
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 6 | 13
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Test type: Superiority; p = 0.11, Chi-squared

4. Secondary Outcome: Percent of Participants With no Significant Nausea in Acute Phase
Description: Reported as acute [chemotherapy days]. All assessment with all VAS < 25 mm on days of chemotherapy
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 33 | 39
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Test type: Superiority; p = 0.28, Chi-squared

5. Secondary Outcome: Percent of Participants With no Significant Nausea in Delayed Phase
Description: Reported for delayed [5 days after chemotherapy administration] All assessment with all VAS < 25 mm
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 16 | 34
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Test type: Superiority; p = 0.002, Chi-squared

6. Secondary Outcome: Percent of Patients With no Nausea in Overall Assessment Period
Description: No nausea (all VAS <5 mm) in overall assessment period (days of chemotherapy plus five days after)
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 6 | 18
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Test type: Superiority; p = 0.006, Chi-squared

7. Secondary Outcome: Percent of Patients With Complete Response in Acute Phase
Description: Complete response (no emesis and no more than minimal nausea, defined as < 25 mm on a 100 mm visual analog scale [VAS]) in acute phase (days of chemotherapy)
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 31 | 39
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Test type: Superiority; p = 0.13, Chi-squared

8. Secondary Outcome: Percent of Patients With Complete Response in Delayed Phase
Description: Complete response (no emesis and no more than minimal nausea, defined as < 25 mm on a 100 mm visual analog scale [VAS]) in delayed phase (5 days after chemotherapy)
Time Frame: Until study completion; estimated 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
Number analyzed (Participants) | 50 | 51
Participants | 15 | 31
Statistical Analysis 1: Comparison: Triplet Therapy Plus Placebo vs Triplet Therapy Plus Olanzapine; Test type: Superiority; p = 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious, and other (non-serious) adverse events were not monitored/assessed during this study. Adverse events were reported only via quantification of number of subjects who withdrew from study for potential adverse events (by patient report or investigator discretion). The time frame in which withdrawal from study was monitored for each patient was the duration of active study period (chemotherapy plus five days after).
Description: All-cause mortality, serious, and other (non-serious) adverse events were not monitored/assessed.
  Adverse events were monitored only by quantifying number of subjects who withdrew from study for potential adverse events (by patient report or investigator discretion).
Arm/Group | Triplet Therapy Plus Placebo | Triplet Therapy Plus Olanzapine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/50 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triplet Therapy Plus Placebo (N=50) | Triplet Therapy Plus Olanzapine (N=51)
Withdrawal From Study (General disorders) | 3 (3) | 0 (0) — Patient or physician request to withdrawal from study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT02635984/Prot_SAP_000.pdf